CLINICAL TRIAL: NCT01107795
Title: Prospective Study to Evaluate Outcomes From Transoral Base of Tongue Resection for Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: Prospective Study to Evaluate Outcomes From Transoral BOT Resection for OSAHS
Status: Terminated | Type: Observational
Why Stopped: Participant attrition before final follow-up visit was greater than anticipated.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kirk P. Withrow, MD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F091104002
Record Dates: First submitted 2010-04-08; First posted 2010-04-21 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transoral Robotic Surgery — Base of tongue resection with transoral robotic-assisted surgery (TORS).

SUMMARY:
This is a prospective observational study that will collect outcome data for patients who choose to undergo transoral tongue base operations for Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)as part of their standard of care treatment. This is a data collection study only and does not provide for evaluations or treatment of OSAHS.

DETAILED DESCRIPTION:
Obstructive sleep apnea hypopnea syndrome (OSAHS) is a major public health problem, and studies suggest that the incidence of OSAHS may be even higher than estimated. Transoral base of tongue resections are commonly preformed to improve symptoms in OSAHS, but among surgeons there is not yet consensus as to the best tongue base operation. The difficulty in treating the tongue base is illustrated by the abundance of available procedures - including genioglossus advancement, hyoid advancement, tongue base suspension, radiofrequency treatment, transoral midline glossesctomy, submucosal coblation-assisted tongue base resection and recently; transoral robotic-assisted surgery (TORS) for base of tongue (BOT) resection. We will evaluate TORS BOT resection for use in OSAHS by assessing pre- and post-operative OSAHS scores and comparing them to historical data for alternative BOT operations.

Though routine, BOT resection may result in significant post-operative pain leading to dysphagia. In certain patients, major complications such as aspiration pneumonia, malnutrition and dehydration can occur as a result. Thus, reducing post-operative dysphagia is critical to improving patient outcomes and limiting complication-associated hospital admissions. Several studies have addressed the management of post-operative dysphagia, but none have evaluated TORS BOT resections in OSAHS. Additionally, TORS BOT resections for malignant neoplasms have been previously shownto be safe and feasible. An outcome analysis of TORS BOT resections for OSAHS may therefore yield recommendations for reducing patient morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with documented OSAHS who is scheduled for tongue base resection at UAB
2. Age > 18
3. Patients must sign informed consent

Exclusion Criteria:

1. Psychological condition that renders the patient unable to understand the informed consent
2. Any situation or condition that will interfere with adherence to study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who choose to undergo transoral robotic assisted tongue base operations for Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS).
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Withrow, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transoral BOT: Participants who received transoral base of tongue surgery as treatment for OASHS.
Period: Overall Study
Arm/Group | Transoral BOT
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transoral BOT
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
Number of Participants Stratified by Apnea Hypopnea Index (AHI) score [Number; unit: participants] — The Apnea Hypopnea Index (AHI) score is the number of apnea and hypopnea events per hour, as recorded during a sleep study. A score from 0 to 14.99 denotes mild sleep apnea; 15 to 29.99 is moderate sleep apnea, while a score of 30 and above is considered severe sleep apnea. Population: Participants with no recorded AHI score were considered eligible for surgery based on the RDI (Respiratory Disturbance Index) score. There is no way to convert an RDI score to an AHI score without access to the original sleep study data, as RDI takes into account all respiratory-effort related arousals.
  participants
    Mild apnea (AHI score of 0 to 14.99) | 8
    Moderate apnea (AHI score of 15 to 29.99) | 5
    Severe apnea (AHI score of 30 or higher) | 17
    no recorded AHI score available | 11

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Apnea Hypopnea Index (AHI) Score
Description: Improvement in Apnea Hypopnea Index (AHI) score, as measured by a polysomnogram sleep study. The AHI score is the number of apnea events per hour, with a lower score indicating mild sleep apnea and a higher score indicating severe sleep apnea. An improved AHI score would be a lower score at 6 months than at 3 months and baseline.
Time Frame: Baseline, 3 months, 6 months
Population: Participant attrition rate was very high; no data were collected.
Arm/Group | Transoral BOT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Transoral BOT
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 4/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transoral BOT (N=41)
syncope (Nervous system disorders) | 1
laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transoral BOT (N=41)
pain (General disorders) | 2
postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
aspiration (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2012-01-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT01107795/Prot_000.pdf